CLINICAL TRIAL: NCT02147548
Title: Evaluation of the Effects of Etifoxine 100 mg and Lorazepam 2 mg on Vigilance and Cognitive Functions in the Elderly. A Monocentric, Randomized, Cross-over, Double-blind Clinical Study Versus Placebo
Brief Title: Evaluation of the Effects of Etifoxine 100 mg and Lorazepam 2 mg on Vigilance and Cognitive Functions in the Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocodex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ETILANCE - ETI 175; NCT02143895 (obsolete NCT alias)
Record Dates: First submitted 2014-05-22; First posted 2014-05-26 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — etifoxine; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- etifoxine (Anxiolytic) (Experimental): etifoxine, 100 mg, a single oral intake
  Interventions: Drug: etifoxine
- lorazepam (Active Comparator): lorazepam, 2 mg, a single oral intake
  Interventions: Drug: lorazepam
- Placebo (Placebo Comparator): 2 capsules of Placebo, a single oral intake
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: etifoxine
  Arms: etifoxine (Anxiolytic)
Drug: lorazepam
  Arms: lorazepam
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of etifoxine (an anxiolytic) compared to lorazepam (a benzodiazepine anxiolytic) on vigilance and cognitive functions in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged from 65 to 75 years
* Right-handed subject (Edinburgh Handedness inventory)
* Subject having signed the consent form
* Subject having agreed to be listed on the French National Healthy Volunteers database
* Subject affiliated or beneficiary to French social insurance

Exclusion Criteria:

* Subject presenting a neurological or psychiatric disease notably cognitive, progressing
* Anxious subject (Hamilton score > 7 and/or Spielberger score > 51 for a man or > 61 for a woman)
* Left-handed subject (Edinburgh Handedness inventory)
* Subject presenting a not corrected visual disease or a motor function disease that could interfere with tests realization
* Smoker
* Subject taking one or more psychotropics or apparent products
* Subject having taken, during the previous month, one or more drugs that could interfere with study drugs metabolism
* Subject drinking too much coffee or tea (> 4 cups per day) or alcohol (>½ liter of wine or equivalent per day)
* Subject presenting contra-indication to one of the drugs used in the study
* Subject with past history of intolerance to drugs used in the study
* Subject not capable to use the CANTAB cognitive evaluation system
* Subject which may not be able to participate to the whole study
* Subject under tutelage or guardianship
* Subject not able to well-understand French and so to understand cognitive tests
* Subject not capable to swallow capsules
* Subject participating to another study or in exclusion period (3 months after a previous trial).

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Reaction time (RTI) of Cambridge Neuropsychological Test Automated Batteries (CANTAB) | 2 hours after the study treatment intake

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Investigation Clinique, CIC 1403 INSERM/CHRU, Lille, France

REFERENCES:
- [Derived] Deplanque D, Machuron F, Waucquier N, Jozefowicz E, Duhem S, Somers S, Colin O, Duhamel A, Bordet R. Etifoxine impairs neither alertness nor cognitive functions of the elderly: A randomized, double-blind, placebo-controlled crossover study. Eur Neuropsychopharmacol. 2018 Aug;28(8):925-932. doi: 10.1016/j.euroneuro.2018.05.011. Epub 2018 Jun 29. PMID 30135030